CLINICAL TRIAL: NCT01674439
Title: Randomized Controlled Clinical Trial of Fat Grafts Supplemented With Adipose-derived Regenerative Cells for Facial Soft Tissue Augmentation in Patients With Craniofacial Microsomia.
Brief Title: Clinical Trial of Fat Grafts Supplemented With Adipose-derived Regenerative Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Y. S. Tanikawa, MD, Assistant Physician, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1069/08; CEPID-FAPESP 98/14254-2 (Other Grant/Funding Number: CEPID-FAPESP 98/14254-2)
Record Dates: First submitted 2012-08-22; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Craniofacial Microsomia
Keywords: Adipose-derived regenerative cells; Cell therapy; Autologous fat transfer; Tissue engineering; Craniofacial microsomia
MeSH Terms: conditions — Goldenhar Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- With supplementation of ADRC (Experimental): Fat graft with supplementation of ADRC
  Interventions: Procedure: Supplementation of ADRC
- Without supplementation of ADRC (Active Comparator): Fat grafts without supplementation of ADRC
  Interventions: Procedure: Without supplementation of ADRC

INTERVENTIONS:
Procedure: Supplementation of ADRC — Isolation of ADRC from half of the aspirated fat and supplementation of the fat grafts with these cells
  Other Names: Cell-assisted lipotransfer
  Arms: With supplementation of ADRC
Procedure: Without supplementation of ADRC — Standard fat graft preparation
  Other Names: Structural fat grafting
  Arms: Without supplementation of ADRC

SUMMARY:
Although first reports of the clinical use of adipose-derived regenerative cells (ADRC) suggest that this approach may be feasible and effective for soft tissue augmentation, there is a lack of randomized, controlled clinical trials in the literature. Hence, this study aimed to investigate whether a novel protocol for isolation of ADRC and their use in combination with fat tissue improve the long-term retention of the grafts in patients with craniofacial microsomia.

DETAILED DESCRIPTION:
To overcome problems associated with fat grafting, such as unpredictable clinical results and a low rate of graft survival, many innovative efforts and refinements of surgical techniques have been reported. For example, condensation of living tissue and removal of unnecessary components have been performed by centrifugation, filtration or gravity sedimentation; external mechanical force has been used to expand the recipient tissue as well as the overlying skin envelope; and a recent experimental study has suggested that repeated local injections of erythropoietin might enhance retention of grafted fat.

Based on the finding that aspirated fat tissue contains a much smaller number of adipose-derived regenerative cells (ADRC) compared with intact tissue and that these cells play pivotal roles in the adipose tissue remodeling after lipoinjection, the supplementation of fat grafts with stromal vascular fraction isolated from adipose portion of liposuction aspirates has been proposed as a method to compensate its relative deficiency of ADRC.

In the literature, there are at least three experimental studies demonstrating that supplementation of adipose progenitor cells enhances the volume or weight of surviving adipose tissue, and first reports of the clinical use of ADRC suggest that this approach may be feasible and effective for soft tissue augmentation.

However, since these studies represent level of evidence IV, which correspond to the publication of case series, there is a lack of randomized, controlled clinical trials comparing this method to current standard techniques.

Hence, this study aimed to fill this gap by investigating whether a novel protocol for isolation of ADRC and their use in combination with fat tissue improve the long-term retention of the grafts in patients with craniofacial microsomia.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral craniofacial microsomia
* 10 to 35 years old
* Phenotype (M0, M1 or M2) and (S1 or S2) according to the OMENS-PLUS classification

Exclusion Criteria:

* Previous soft tissue surgery
* Absence of fat donor site

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Graft volume retention | 6 months postoperative
  Graft volume retention evaluated by CT-scan performed at the preoperative period and at 6-months postoperative

SECONDARY OUTCOMES:
Number of viable cells before and after the supplementation of the grafts | immediate postoperative
  Number of viable cells in adipose tissue evaluated by trypan blue method immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Y Tanikawa, MD, Principal Investigator — Division of Plastic and Reconstructive Surgery, University of São Paulo School of Medicine
Locations (1):
- Division of Plastic and Reconstructive Surgery, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Yoshimura K, Sato K, Aoi N, Kurita M, Hirohi T, Harii K. Cell-assisted lipotransfer for cosmetic breast augmentation: supportive use of adipose-derived stem/stromal cells. Aesthetic Plast Surg. 2008 Jan;32(1):48-55; discussion 56-7. doi: 10.1007/s00266-007-9019-4. Epub 2007 Sep 1. PMID 17763894
- [Result] Yoshimura K, Sato K, Aoi N, Kurita M, Inoue K, Suga H, Eto H, Kato H, Hirohi T, Harii K. Cell-assisted lipotransfer for facial lipoatrophy: efficacy of clinical use of adipose-derived stem cells. Dermatol Surg. 2008 Sep;34(9):1178-85. doi: 10.1111/j.1524-4725.2008.34256.x. Epub 2008 May 29. PMID 18513295
- [Result] Yoshimura K, Asano Y, Aoi N, Kurita M, Oshima Y, Sato K, Inoue K, Suga H, Eto H, Kato H, Harii K. Progenitor-enriched adipose tissue transplantation as rescue for breast implant complications. Breast J. 2010 Mar-Apr;16(2):169-75. doi: 10.1111/j.1524-4741.2009.00873.x. Epub 2009 Nov 12. PMID 19912236
- [Result] Yoshimura K, Eto H, Kato H, Doi K, Aoi N. In vivo manipulation of stem cells for adipose tissue repair/reconstruction. Regen Med. 2011 Nov;6(6 Suppl):33-41. doi: 10.2217/rme.11.62. PMID 21999260